CLINICAL TRIAL: NCT02949713
Title: Feasibility and Effects of Mobile Phone Text Messaging Plus Motivational Interviewing Versus Usual Care in Promotion of Breastfeeding Among HIV-infected Women in South Africa: A Randomized, Parallel Group, Controlled Pilot Trial
Brief Title: Text Messaging Plus Motivational Interviewing in Promotion of Breastfeeding Among HIV-infected Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Stellenbosch (Other)
Collaborators: McMaster University (Other); University of British Columbia (Other)
Responsible Party: Principal Investigator, Moleen Zunza, Dr, University of Stellenbosch
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: N16/09/11
Record Dates: First submitted 2016-10-26; First posted 2016-10-31 (Estimated); Last update posted 2023-09-26 (Actual); Status verified 2023-09

CONDITIONS: HIV Infections; Breast Feeding
Keywords: HIV; infant feeding; mHealth; behavioural intervention
MeSH Terms: conditions — HIV Infections; Breast Feeding | interventions — Motivational Interviewing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Text messaging-motivational interviewing (Experimental): Every Monday morning, a text message (SMS) will be sent to participants in the intervention group encouraging participants to continue breastfeeding, and inquire if participants have any problems breastfeeding their infants. Participants will be asked to respond within 48 hours, indicating that they either do not have a problem or they have a problem and require help. In addition to text messaging, participants will have motivational interviews post-delivery at weeks 2, 6, and 10. Motivational interviews will explore and support the participant's commitment to continue breastfeeding.
  Interventions: Behavioral: Text messaging-motivational interviewing
- Usual standard of care (No Intervention): Usual standard of care

INTERVENTIONS:
Behavioral: Text messaging-motivational interviewing — Interactive weekly mobile phone text messaging plus prospective motivational interviews
  Other Names: mobile phone text messaging; motivational interviewing
  Arms: Text messaging-motivational interviewing

SUMMARY:
The primary aim of this study is to find out whether it is feasible to conduct a larger study looking at the effect of mobile phone text messaging added to motivational interviewing on number of participants invited to the study who consented to participate and the number with complete evaluation of infant feeding practices at all study visits.

Secondary aim: In HIV-infected women initiating breastfeeding after giving birth, does interactive weekly mobile phone text messaging plus motivational interviewing versus usual care, improve self-reported adherence to exclusive or any breastfeeding 6 months post-delivery and to determine the number of women remaining in the group they were assigned until end of study or lost to follow-up (protocol adherence).

DETAILED DESCRIPTION:
Breastfeeding reduces the risks of dying from infections and is currently recommended as the most beneficial feeding option for infants born to HIV-infected women in low-resourced settings. This recommendation contradicts previous recommendations to avoid breastfeeding to prevent mother-to-child transmission of HIV. South Africa, a high HIV prevalent country, recently phased out access to free formula milk in the public sector in support of breastfeeding for HIV-infected women. The investigators previously found that few HIV-infected South African women choose breastfeeding and among those who did, many stop breastfeeding early. This study involves text messaging breastfeeding advice encouraging women to exclusively breastfeed, and inquire if they have any breastfeeding related problems, and motivational interviews exploring and supporting woman's commitment to continue breastfeeding.Participants meeting inclusion criteria who consent participation will be enrolled by a research nurse and immediately randomly assigned to text messaging plus motivational interviewing group or usual standard of care group.

The investigators propose a randomized, parallel group, standard of care-controlled pilot trial which will be conducted among HIV-infected women of low socio-economic background, giving birth at a primary healthcare clinic in Cape Town, South Africa. The pilot trial will assess the feasibility of conducting a larger trial on communication and support approaches that may improve HIV-infected woman's adherence to exclusive and continued breastfeeding.

ELIGIBILITY:
Inclusion Criteria:

* Women living with HIV
* initiated breastfeeding within 24 hours of giving normal birth
* on ART
* 18 years or older
* ownership of a mobile phone
* infants judged to be in good health who are discharged soon after delivery

Exclusion Criteria:

* initiating both breastfeeding and formula feeding or formula feeding within 24 hours of giving birth.
* gave birth to more than one infant
* birth weight < 2500
* gestational age < 36 weeks

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2019-05-02 (Actual); Primary Completion 2020-08-13 (Actual); Study Completion 2020-08-13 (Actual)

PRIMARY OUTCOMES:
Number of participants invited to the study who consented to participate. | 6 month post randomization
  Number of participants invited to the study who consented to participate.
Number of participants with complete evaluation of infant feeding practices at all study visits | 6 month post randomization
  Number of participants with complete evaluation of infant feeding practices at all study visits as assessed by infant feeding questionnaire.

SECONDARY OUTCOMES:
Number of participants remaining in the group they were assigned until end of study or lost to follow-up (protocol adherence). | 6 month
  Number of participants remaining in the group they were assigned until end of study or lost to follow-up (protocol adherence).
Number of participants who are exclusively breastfeeding | 6 month post randomization
  Number of participants who report giving only breast milk and no other liquids or solid based foods to their infants as assessed by the infant feeding questionnaire
Number of participants who are breastfeeding | 6 month post randomization
  Number of participants who report giving breast milk and other liquids or solid based foods to their infants as assessed by the infant feeding questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Moleen Zunza, Principal Investigator — University of Stellenbosch; Taryn Young, Study Chair — University of Stellenbosch; Mark F Cotton, Study Chair — University of Stellenbosch; Lehana Thabane, Study Chair — McMaster University
Locations (1):
- Moleen Zunza, Cape Town, Western Cape, South Africa

IPD SHARING:
Plan to Share IPD: Yes
The IPD will be available from the corresponding author on reasonable request
Supporting Information: Study Protocol, ICF
Time Frame: Data will be available until year 2035.
Access Criteria: Investigators conducting maternal-child health studies with appropriate institutional review board approvals for any additional pooled analyses, will have access to the anonymized and de-identified individual participant data, from the corresponding author on reasonable request.

REFERENCES:
- [Derived] Zunza M, Young T, Cotton M, Slogrove A, Mbuagbaw L, Kuhn L, Thabane L. Evaluating interactive weekly mobile phone text messaging plus motivational interviewing for breastfeeding promotion among women living with HIV, giving normal birth at a primary healthcare facility in South Africa: a feasibility randomised controlled trial. BMJ Open. 2023 Oct 10;13(10):e073385. doi: 10.1136/bmjopen-2023-073385. PMID 37816561
- [Derived] Zunza M, Cotton MF, Mbuagbaw L, Lester R, Thabane L. Interactive weekly mobile phone text messaging plus motivational interviewing in promotion of breastfeeding among women living with HIV in South Africa: study protocol for a randomized controlled trial. Trials. 2017 Jul 17;18(1):331. doi: 10.1186/s13063-017-2079-0. PMID 28716146